CLINICAL TRIAL: NCT02010294
Title: Invasive Group A Streptococcus (GAS) Infection in Children: Bacterial Virulence Factors and Detection of Host Immunological and/or Genetic Factors of Predisposition to Infections
Acronym: StreptoPedia
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: P120136
Record Dates: First submitted 2013-11-21; First posted 2013-12-12 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2018-02

CONDITIONS: Invasive GAS Infection
Keywords: Invasive GAS infection; emm genotypes; Bacterial virulence factors; Mendelian susceptibility to infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Children hospitalized for invasive GAS infection: Children hospitalized for invasive GAS infection
  Interventions: Genetic: DNA samples, GAS strains
- Children with non-invasive infection: Children with non-invasive infection such as pharyngitis, tonsillitis, proctitis or skin infection diagnosed by a positive test for rapid diagnosis of GAS performed at the site of infection with a positive GAS culture
  Interventions: Genetic: DNA samples, GAS strains

INTERVENTIONS:
Genetic: DNA samples, GAS strains — DNA samples,GAS strains

SUMMARY:
The main objective of the study is to characterize the virulence factors of SGA and identify immunological and / or genetic factors predisposing to infections in children hospitalized with invasive GAS infection.

DETAILED DESCRIPTION:
The group A streptococcus (GAS) or Streptococcus pyogenes is a strictly human pathogen , which can cause a wide variety of infections. These range from a simple asymptomatic carriage up to 20 % of children , or minor illnesses such as sore throat or impetigo, to severe conditions such as necrotizing fasciitis and toxic shock syndrome .

The pathophysiological mechanisms of invasive GAS infections are poorly understood. These mechanisms could involve not only virulence factors of the bacterium ( M protein determines the emm genotype , but also super- antigenic exotoxins SpeA , Spe C, Ssa, Sme z or other virulence genes , SilC , ... Sic ), but also in some cases, factors associated with host immunity in particular in the absence of risk factors for invasive skin infection such as cutaneous effraction ( wound , burn , chicken pox ) , corticosteroids or other immunosuppressive therapy and recent surgery .

The investigators assume that in some invasive GAS infections, especially in children without risk factors, Mendelian susceptibility to infection may be involved . This hypothesis could be tested by studying the molecular characteristics of strains isolated SGA and innate and adaptive immunity in children hospitalised for invasive GAS infection with or without identified risk factors for infection.

This study could not only lead to a better understanding of the pathophysiological mechanisms of invasive GAS infections but also to detect in children who underwent invasive GAS genetic susceptibility to infections requiring specific care . Finally, it could also identify specific strains of SGA or molecular profiles, whose detection in practice, lead to a suspicion of hereditary immune deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 1 month to <15 years at the time of inclusion
* Group 1 : Children hospitalized for invasive GAS infection

  * Subgroup 1A ( N = 75 ): Children with invasive infection without known risk factor .
  * Subgroup 1B (N = 75) : Children with invasive infection with known risk factor .

GAS Invasive infections are defined by:

a) Proved infection : Bacteriological isolation of S. pyogenes from a liquid or a normally sterile site, except from a blister of a simple erysipelas, without necrosis . This is sometimes associated with a shock with multiorgan failure (streptococcal toxic shock syndrome ( STSS )) b ) Probable infection :

1. . Bacteriological isolation of S. pyogenes from a normally non-sterile site ( eg skin, upper respiratory tract ) associated with extensive soft tissue necrosis
2. . Bacteriological isolation of S. pyogenes a site or a biological sample usually non-sterile ( eg skin , upper respiratory tract ) associated with a evocative shock syndrome STSS and no other cause found .

Contributing factors for invasive infection are defined by:

cutaneous effraction (wounds , burn , chicken pox ), the use of corticosteroids or other treatment, immunosuppressive and recent surgery

• Group 2: non-invasive infection such as pharyngitis , tonsillitis, proctitis or skin infection diagnosed by a positive test for rapid diagnosis of GAS performed at the site of infection with a positive GAS culture.

Exclusion Criteria:

* Group 1: Children with a known immune deficiency unrelated to the risk factors described above.
* Group 2: Children with a known immune deficiency.

Ages: 1 Month to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children hospitalized for invasive or non invasive GAS infection
Sampling Method: Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2014-02-10 (Actual); Primary Completion 2018-02-10 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
virulence factors of GAS | up to 3 years
  characterize the virulence factors of GAS

SECONDARY OUTCOMES:
Assess the frequency and type of hereditary immune deficiency or Mendelian susceptibility to infections associated with invasive GAS infections in children without risk factors | up to 3 years
  frequency and type of hereditary immune deficiency or Mendelian susceptibility to infections associated with invasive GAS infections
describe and compare the GAS emm genotypes and virulence factors with the profiles of strains isolated with invasive GAS infection with known risk factors and with the profile of strains isolated with a non-invasive GAS infections | up to 3 years
  describe and compare the GAS emm genotypes and virulence factors profile of GAS associated with an inherited immune deficiency, or a Mendelian susceptibility to infection, with the profiles of strains isolated in children with invasive GAS infection with known risk factors (use of steroids, varicella, wounds…) and with the profile of strains isolated in children with a non-invasive GAS infections
compare GAS emm genotypes and profiles of virulence strains responsible for invasive SGA infections with strains causing noninvasive infections | up to 3 years
  compare GAS emm genotypes and profiles of virulence strains responsible for invasive SGA infections with strains causing noninvasive infections

CONTACTS AND LOCATIONS:
Overall Officials: Albert FAYE, MD, PhD, Principal Investigator — APHP
Locations (1):
- Robert Debré Hospital, Paris, France